CLINICAL TRIAL: NCT02229448
Title: A Survey of Patients With Elevated Serum IGG4 With Unknown IGG4-related Disease to Whom Biopsy and Performance of Subsequent Specific Staining for Clinical, Laboratory and Pathologic Correlation.
Brief Title: Retrospective Study for Diagnosis of Undetected IgG4 Related Diseases in Patients With High Serum IgG4 Levels.
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, yair levy, Meir Medical Center, Meir Medical Center
Other Study IDs: IgG4-RD diagnosis
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2014-08

CONDITIONS: Undiagnosed IgG4 Related Diseases
Keywords: Immunoglobulin G; focus; study; detect; patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IgG4 UKN diagnosis: who ever been found with IgG4 sub class in blood sample or in his byposy

SUMMARY:
Immunoglobulin G4-related disease (IgG4-RD) is an increasingly recognized syndrome of unknown etiology comprised of a collection of disorders that share specific pathologic, serologic, and clinical features.

Histopathological analysis of biopsy specimens remains the cornerstone in the diagnosis of IgG4- related disease. Elevated concentrations of IgG4 in tissue and serum are helpful in diagnosing IgG4-related disease, but neither one is a specific diagnostic marker. Correlation with specific histopathological findings is essential, regardless of the serum IgG4 concentration, the number of IgG4-positive plasma cells in tissue, or the ratio of IgG4 to IgG in tissue. Misdiagnoses of IgG4-related disease are increasingly common because of excessive emphasis on moderate elevations of serum IgG4 concentration and overreliance on the finding of IgG4-positive plasma cells in tissue.

DETAILED DESCRIPTION:
IgG4 is a unique antibody in both structure and function. This molecule accounts for less than 5% of the total IgG in healthy persons and is the least abundant IgG subclass. In contrast to IgG1, IgG2, and IgG3, serum IgG4 concentrations among ostensibly healthy people vary by a factor of more than 100 (normal range, 0.01 to 1.4 mg per milliliter), but IgG4 concentrations within individual persons are generally stable.

Immunoglobulin G4-related disease (IgG4-RD) is an increasingly recognized syndrome of unknown etiology comprised of a collection of disorders that share specific pathologic, serologic, and clinical features.

These different conditions were previously thought to be unrelated [2-4]. The commonly shared features include tumor-like swelling of involved organs, a lymphoplasmacytic infiltrate enriched in IgG4-positive plasma cells, and variable degrees of fibrosis that has a characteristic "storiform" pattern. In addition, elevated serum concentrations of IgG4 are found in 60 to 70 percent of patients with IgG4-RD.

Two major presentations of this condition, which often affects more than one organ, are type 1 autoimmune pancreatitis (IgG4-related pancreatitis) and salivary gland disease; the later may present as salivary gland enlargement or as sclerosing sialadenitis (formerly termed "Mikulicz disease" and Küttner's tumor, respectively). These conditions often resemble Sjögren's syndrome but are pathophysiologically distinct from this disorder. The preferred name for the overall condition is IgG4-related disease.

The presence of IgG4-bearing plasma cells is required for a diagnosis of IgG4- related disease, but IgG4-positive cells are found in a wide variety of inflammatory infiltrates, and the detection of substantial numbers of IgG4- positive plasma cells is therefore not diagnostic of IgG4-related disease.

Tissues from patients with IgG4-related disease show diffuse infiltrates of IgG4-bearing plasma cells, in contrast to the focal aggregates of IgG4-bearing cells that are detected in most other inflammatory mimickers of this condition. A diffuse plasma-cell infiltrate with more than 30 IgG4-positive cells per high power field and a ratio of IgG4 to IgG that is higher than 50% provides compelling evidence of IgG4-related disease.

The study will examine the clinical data from the computerized database of Meir Hospital for patient with unknown IGG4-related disease with high serum levels of IGG4 that were admitted for hospitalization for any reason in a period of 14 years, from January 2000 to June 2014.

Since biopsy has proven to be the hallmark in diagnosing IGG4 RD, we decided to complete the investigation in a pool of patients to whom high IGG4 serum levels where confirmed and to whom biopsies from any suitable tissue where obtained for other reasons than IGG4 RD and then to perform specific staining for IGG4 to those samples, by sending them back to the pathology service at our hospital.

Furthermore clinical and other laboratory features of each positive patient will then be correlated from the history of admission of each patient.

ELIGIBILITY:
Inclusion Criteria:

* All patients that where admitted during the period of January 2000 to June 2014 at MEIR HOSPITAL KFAR SAVA, with at least one result of a high serum level of IGG4 according to the accepted normal range in our laboratory (more than 100mg/dL) and to whom biopsy of a suitable tissue was obtained for other reasons than IGG4 Related Diseases.
* Both genders will be included.
* Patients of all ages.

Exclusion Criteria:

* Patients who have already been diagnosed with IGG4-Related Diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that where admitted during the period of January 2000 to June 2014 at MEIR HOSPITAL- KFAR SABA from all ages, from all parts of Israel, all races will be included, from both genders.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
serum level of IGG4 | 6 months
  Taken from a computerized database

SECONDARY OUTCOMES:
specific staining for IGG4 to biopsy samples | six months
  took from biposy that save for clinical trails

CONTACTS AND LOCATIONS:
Overall Officials: Yair Levy, MD, Principal Investigator — Meir Medical Center; Shalabi Khaled, Study Chair — Meir Medical Center; Evgeny Edelshtein, MD, Study Chair — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel